CLINICAL TRIAL: NCT04432116
Title: EEG and Behavioural Correlates of Virtual Reality Treatment of Environmental Zeitgebers in Schizophrenia and Bipolar Disorder
Brief Title: Time and Virtual Reality in Schizophrenia and Bipolar Disorder
Acronym: VirtualTimes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: C19-48
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: All interventions are applied to each participant
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- virtual reality 1 (Experimental): the subject is in a virtual room and is asked to emit a retrospective time duration judgement at the end of the session
  Interventions: Behavioral: virtual reality 1
- virtual reality 2 (Experimental): the subject is in a virtual environment mimicking a space ship. The subject is asked to detect targets as fast as possible while the background of the virtual environment is a starfield with standard speed vs. self-determined speed vs. static stars
  Interventions: Behavioral: virtual reality 2
- virtual reality 3 (Experimental): the subject is in a virtual environment mimicking a space ship. The subject is asked to detect targets as fast as possible.Asynchronous distracters vs. synchronous distracters, vs no distracters are displayed while the subjects wait for the target
  Interventions: Behavioral: virtual reality 2

INTERVENTIONS:
Behavioral: virtual reality 1 — the subject is in a virtual waiting room, there is no other intervention. The principle of this intervention is to make the subject wait with as little interfering events as possible
  Arms: virtual reality 1
Behavioral: virtual reality 2 — Subjects are in a virtual environment mimicking a space ship. On the screen there is a red light and subjects wait for this red light to become green. They press on a pad each time the red light becomes green
  Other Names: virtual reality 3
  Arms: virtual reality 2; virtual reality 3

SUMMARY:
Patients with bipolar disorders report an acceleration or slowing of time flow, and patients with schizophrenic spectrum disorders a time fragmentation. These disorders would be linked to disorders of the sense of self. Assessing these time-related disorders could help to better predict psychotic conversion in vulnerable subjects. In this protocol, the investigators wish to develop playful methods for the evaluation of alterations in the passage of time, based on the use of virtual reality. The protocol will be tested in stabilized but chronic bipolar or schizophrenic patients, vs. healthy subjects matched on age, sex, and study level. The protocol will include two experimental sessions. It will begin with a waiting room-like session, at the end of which the subject will be asked to retrospectively estimate the time that will have passed. The games that will follow will all be based on the principle of temporal waiting. A first signal will indicate the start of the trial, and a target will be presented at varying times after this first signal. The later the target is presented, the more the subject expects and prepare for the target, and the faster he or she is. This time delay is measured by the subject's response (response time, error rate, eye fixation), but also by electrical signals measured by electroencephalography (EEG). The two experimental sessions will include several temporal manipulations during these tasks, intended to highlight alterations in the time flow in patients compared to controls. In one of the sessions, a starfield will be presented and the speed of the stars in the starfield will be manipulated, as a proxy for the speed of the environment. In one condition, the speed of the object will be average, and in the other the speed will be self-adjusted by the subject. In a control condition, the speed of the object will be zero. In the other experimental session, distractors will be presented during the waiting phase of the target. They will be presented either simultaneously or asynchronously. In one control condition the distractors will be absent. In both sessions it will be examined how the behavioral and EEG cues are affected by the manipulations. A double dissociation is expected, with greater disturbance in patients with bipolar disorder when standard movement is used, whereas patients with schizophrenia should be disturbed mainly when asynchronous distractors are presented.

ELIGIBILITY:
Inclusion Criteria:

* - Participant, male or female, between 18 and 60 years old
* Subject affiliated to a social health insurance scheme (beneficiary or entitled person)
* Subject who has dated and signed an informed consent form
* For a woman of childbearing age, negative pregnancy test and effective contraception throughout the study
* A patient under guardianship, whose guardian has dated and signed a consent, as well as the patient if able.
* A patient under guardianship, whose consent has been obtained, if necessary, by the guardian or with the assistance of the guardian, prior to the commencement of any trial-related procedures.

Patients only:

* Patients with psychotic disorders (schizophrenia-like): Patients with diagnostic criteria for schizophrenia as defined by the DSM V (American Psychiatric Association, 2015).
* Patients with Bipolar Disorder: A patient with diagnostic criteria for bipolar disorder as defined by the DSM V (American Psychiatric Association, 2015).

Exclusion Criteria:

* Substance Use Disorders (as defined by DSM-V)
* Intake of benzodiazepines (in the period before inclusion, for a duration equivalent to 5 half-lives of the product), cannabis (in the 2 months before inclusion) or hallucinogenic substances (in the period before inclusion, for a duration equivalent to 5 half-lives of the product).
* A neurological pathology or sequelae
* Attention Deficit Hyperactivity Disorder (ADHD)
* Borderline personality disorder
* Disabling sensory impairment, including visual acuity (corrected, if applicable) < 0.8 (due to the use of visual aids) (Freiburg Vision Test, Bach 1996)
* Person deprived of liberty or under the safeguard of justice
* Pregnant, parturient or breastfeeding women
* Subject in a period of exclusion defined by another clinical study.

Healthy volunteers only:

History of major neurological or psychiatric illness with ongoing psychotropic medication (i.e., antidepressant, thyroid regulator, antipsychotic, benzodiazepine or hypnotic).

Patients only:

Only patients treated with neuroleptics, whether or not combined with an anti-parkinsonian corrector or anti-depressant, will be included. Patients taking benzodiazepines will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
EEG index of time expectation | through study completion, an average of 2 years
  beta oscillations recorded with EEG during the waiting period

SECONDARY OUTCOMES:
retrospective duration | through study completion, an average of 2 years
  Retrospective duration judgement

CONTACTS AND LOCATIONS:
Locations (1):
- Services de Psychiatrie I et II - Pôle de Psychiatrie CHRU Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No